CLINICAL TRIAL: NCT00248456
Title: A Randomised, Double-blind, Active-controlled, Parallel, Multi-center Study to Investigate the Efficacy and Safety of Daivobet® Ointment in Patients With Psoriasis Vulgaris
Brief Title: Efficacy and Safety of Calcipotriol Plus Betamethasone Dipropionate Ointment in Patients With Psoriasis Vulgaris
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EX 0501 CN
Record Dates: First submitted 2005-11-03; First posted 2005-11-04 (Estimated); Last update posted 2025-02-24 (Actual); Status verified 2008-02

CONDITIONS: Psoriasis Vulgaris
MeSH Terms: interventions — calcipotriene

INTERVENTIONS:
Drug: Calcipotriol plus betamethasone dipropionate ointment

SUMMARY:
This study will evaluate the efficacy and safety of calcipotriol plus betamethasone dipropionate ointment compared with calcipotriol ointment in the treatment of patients with psoriasis vulgaris for a duration of 4 weeks. The study will focus on the percentage change of the psoriasis area and severity index (PASI) from baseline to the end of week 4.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of psoriasis vulgaris in a stable condition
* Extent of at least 10% of one or more body regions
* Amenable to topical therapy with maximum of 100 g/week of investigational product

Exclusion Criteria:

* Patients with more than 30% of body surface area involved
* Patients with facial psoriasis who need treatment
* Patients who need treatment of scalp psoriasis with WHO group IV topical corticosteroids, tretinoin or topical vitamin D derivatives
* Patients with unstable forms of psoriasis including guttate, erythrodermic, pustular, or arthritis psoriasis
* Systemic treatment of psoriasis with corticosteroids or other therapy
* Systemic antipsoriatic treatment (e.g. corticosteroids, immunosuppressive drugs, tretinoin, antibiotics, phototherapy or calcium agents) within 4 weeks prior to visit 1; or topical antipsoriatic treatment (e.g. keratolytics, topical corticosteroids, topical vitamin D derivatives, anthralin, crude coal tar, etc) within the previous 2 week period
* Patients with planned exposure to phototherapy that may affect the psoriasis during the study period

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320
Dates: Start 2005-10; Study Completion 2006-02

PRIMARY OUTCOMES:
The percentage change of PASI at the end of week 4 compared with baseline

SECONDARY OUTCOMES:
The change of PASI at the end of week 4 compared with baseline
The change of Dermatology Life Quality Index at the end of week 4 compared with baseline
Physician's Global Assessment at the end of week 4
Patient's assessment by Visual Analogue Scale (VAS) at the end of week 4
The change of individual scores of redness, thickness, and scaliness at the end of week 4 on the target lesion compared with baseline
The change of overall lesion area percentage (scalp and face area excluded) at the end of week 4 compared with baseline

CONTACTS AND LOCATIONS:
Overall Officials: Zheng Zhi Zhong, Professor, Principal Investigator — Fudan University First Hospital, Dermatology Department
Locations (1):
- Fudan University First Hospital, Dermatology Department, Shanghai, China

IPD SHARING:
Plan to Share IPD: No